CLINICAL TRIAL: NCT00962754
Title: Reliability and Utility of Fluid Balance Charting in Neonates Admitted to the Pediatric Ward.
Brief Title: Fluid Balance Study in Sick Neonates
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Princess Amalia Children's Clinic (Other)
Responsible Party: Principal Investigator, Jolita Bekhof, MD, Pediatrician, Princess Amalia Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL26894.075.09
Record Dates: First submitted 2009-08-18; First posted 2009-08-20 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Very Low Birth Weight Infant
Keywords: recording fluid balance; reliability; utility; sick neonate; fluid balance; inpatient; sick

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- physician insight fluid balance (No Intervention): physician has insight in fluid balance chart, this is standard practice
- fluid balance data masked to physician (Experimental): physician no insight in the fluid balance chart
  Interventions: Procedure: physician no insight in the fluid balance chart

INTERVENTIONS:
Procedure: physician no insight in the fluid balance chart — physician had no insight in the fluid balance chart during the first 3 days of admission of the patient when the balance is recorded
  Arms: fluid balance data masked to physician

SUMMARY:
The purpose of this study is to determine if routinely recording fluid balance in sick neonates admitted to the pediatric ward is reliable and useful. The investigators' hypothesis is that it is not useful and reliable.

DETAILED DESCRIPTION:
Fluid balance charts are commonly used, in the Netherlands, to assess patient fluid volume status. Some disadvantages of recording fluid intake and output are that it is time-consuming and complex. If it would give reliable and accurate information about the fluid volume status there would be a good reason for all this effort. In the few researches that have investigated this subject a low correlation has been found between the fluid balance and the weight changes of an adult patient. Own experience gives reasons to doubt about the reliability of the fluid balance in children, not rarely there is a discrepancy between the fluid balance and the weight measurement. We are interested in the relevance of recording fluid balance in neonates.

ELIGIBILITY:
Inclusion Criteria:

* Sick neonates admitted to the neonatal ward

Exclusion Criteria:

* Admitted elsewhere before admission to the neonatal ward
* Indication for recording fluid balance
* Impossibility to measure the weight every day
* No consent parents

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 170 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Bekhof, pediatrician, Study Director — Princess Amalia Children's Clinic; Y v Asperen, MD, Principal Investigator — University of Groningen
Locations (1):
- Princess Amalia Children's Clinic, Zwolle, Overijssel, Netherlands

REFERENCES:
- [Background] Daffurn K, Hillman KM, Bauman A, Lum M, Crispin C, Ince L. Fluid balance charts: do they measure up? Br J Nurs. 1994 Sep 8-21;3(16):816-20. doi: 10.12968/bjon.1994.3.16.816. PMID 7950261
- [Background] Chung LH, Chong S, French P. The efficiency of fluid balance charting: an evidence-based management project. J Nurs Manag. 2002 Mar;10(2):103-13. doi: 10.1046/j.0966-0429.2001.00296.x. PMID 11882111
- [Background] Wise LC, Mersch J, Racioppi J, Crosier J, Thompson C. Evaluating the reliability and utility of cumulative intake and output. J Nurs Care Qual. 2000 Apr;14(3):37-42. doi: 10.1097/00001786-200004000-00005. PMID 10826233
- [Background] Eastwood GM. Evaluating the reliability of recorded fluid balance to approximate body weight change in patients undergoing cardiac surgery. Heart Lung. 2006 Jan-Feb;35(1):27-33. doi: 10.1016/j.hrtlng.2005.06.001. PMID 16426933
- [Background] Mank A, Semin-Goossens A, Lelie Jv, Bakker P, Vos R. Monitoring hyperhydration during high-dose chemotherapy: body weight or fluid balance? Acta Haematol. 2003;109(4):163-8. doi: 10.1159/000070964. PMID 12853687
- [Background] Pflaum SS. Investigation of intake-output as a means of assessing body fluid balance. Heart Lung. 1979 May-Jun;8(3):495-8. PMID 254670
- [Background] Scales K, Pilsworth J. The importance of fluid balance in clinical practice. Nurs Stand. 2008 Jul 30-Aug 5;22(47):50-7; quiz 58, 60. doi: 10.7748/ns2008.07.22.47.50.c6634. PMID 18777823
- [Derived] Bekhof J, van Asperen Y, Brand PL. Usefulness of the fluid balance: a randomised controlled trial in neonates. J Paediatr Child Health. 2013 Jun;49(6):486-92. doi: 10.1111/jpc.12214. Epub 2013 May 2. PMID 23635344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited upon admission to our neonatal high care ward from June 2009 to March 2010
Groups:
- Physician Insight Fluid Balance: Physician has insight in the fluid balance chart
- Physician no Insight Fluid Balance Chart: physician does not have insight in the fluid balance chart
Period: Overall Study
Arm/Group | Physician Insight Fluid Balance | Physician no Insight Fluid Balance Chart
Started | 86 | 84
Completed | 86 | 84
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Physician Insight Fluid Balance: physician has insight in the fluid balance data
- Physician no Insight Fluid Balance Chart: physician does not have insight in the fluid balance data (fluid balance chart is blinded)
- Total: Total of all reporting groups
Arm/Group | Physician Insight Fluid Balance | Physician no Insight Fluid Balance Chart | Total
Number analyzed (Participants) | 86 | 84 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 86 | 84 | 170
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.01 (0) | 0.01 (0) | 0.01 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 70
  Male | 49 | 51 | 100
Region of Enrollment [Number; unit: participants]
  Netherlands | 86 | 84 | 170

OUTCOME MEASURES:

1. Primary Outcome: Duration of Admission at the Ward in Days
Description: Duration of hospital stay in days or duration of admission at the pediatric ward in days
Time Frame: 1-8 months
Population: intention to treat analysis
Measure: Median (Full Range); unit: number of days
Groups:
- Intervention Group (no Insight in Fluid Balance): physician has no insight in fluid balance chart, ie the fluid balance chart is masked
- Control Group (Insight in Fluid Balance): physician has insight in (full access to) the fluid balance chart data
Arm/Group | Intervention Group (no Insight in Fluid Balance) | Control Group (Insight in Fluid Balance)
Number analyzed (Participants) | 84 | 86
number of days | 9 [2 to 37] | 8 [2 to 27]
Statistical Analysis 1: Comparison: Intervention Group (no Insight in Fluid Balance) vs Control Group (Insight in Fluid Balance); We calculated that 85 patients in each group would give a power in excess of 85% to detect a difference of two days or more in the geometric mean length of hospital stay with a two-sided significance level of 0.05; Test type: Non-Inferiority or Equivalence — non-inferiority since our hypothesis was that there would be no difference in outcome between the intervention and the control group; p < 0.05, t-test, 2 sided — log transformation of mean duration of hospitalization,difference between two groups expressed as ratio of geometric means for duration. 95% confidence intervals calculated using bootstrapping method. correction by linear regression model; Adjusted ratio of geometric means = 1, 95% CI 2-sided [0.81 to 1.19]

2. Secondary Outcome: Use of Diuretics
Description: prescription of diuretic therapy
Time Frame: during days of admission
Measure: Number; unit: participants
Groups:
- Intervention Group (no Insight in Fluid Balance): physician has no insight in the fluid balance chart data (masked)
Arm/Group | Intervention Group (no Insight in Fluid Balance) | Control Group (Insight in Fluid Balance)
Number analyzed (Participants) | 84 | 86
participants | 0 | 0

3. Secondary Outcome: Complications
Description: notifications of complications
Time Frame: duration of admission
Measure: Number; unit: participants
Groups:
- Physician Insight Fluid Balance: Physician has insight (full access to) in the fluid balance chart data
- Physician no Insight Fluid Balance Chart: physician has no insight in the fluid balance data (masked)
Arm/Group | Physician Insight Fluid Balance | Physician no Insight Fluid Balance Chart
Number analyzed (Participants) | 86 | 84
participants | 2 | 5

ADVERSE EVENTS:
Groups:
- Physician Insight Fluid Balance: physician has insight in (full access to) the fluid balance chart data
- Physician no Insight Fluid Balance Chart: Physician has no insight in the fluid balance chart data (masked)
Arm/Group | Physician Insight Fluid Balance | Physician no Insight Fluid Balance Chart
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/84
Other Adverse Events (participants affected / at risk) | 0/86 | 0/84

LIMITATIONS AND CAVEATS:
* lack of a more reliable assessment method of fluid status, for example central venous pressure or body impedance measurements
* moderate disease severity
* unequal distribution of premature infants amongst the study groups

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes